CLINICAL TRIAL: NCT06835400
Title: An Open-Label, Randomized, Two-stage Study to Determine Dose Optimization, Safety, and Noninferiority of Oral Paclitaxel + Encequidar Compared to IV Paclitaxel in Subjects With HER2 Negative Metastatic Breast Cancer
Brief Title: Oral Paclitaxel + Encequidar vs IV Paclitaxel in Treatment of HER2 Negative Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Health Hope Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHP-ORAX-300
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: HHP-ORAX-300 is a Phase 3, open-label, randomized, two-stage dose optimization and noninferiority study.
  The study includes 2 stages: Stage 1 is a dose-optimization design that will select an Oral Paclitaxel + Encequidar regimen to test against IV paclitaxel 80 mg/m2 in a confirmatory Stage 2.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stage 1: Oral Paclitaxel 165 mg/m2 + Encequidar (Experimental): A minimum of 20 subjects per group will be centrally randomized 1:1 to Oral Paclitaxel 165 mg/m2 + Encequidar 3 weeks of a 4-week cycle (3/4) or Oral Paclitaxel 205 mg/m2 (3/4) + Encequidar.
  Interventions: Drug: Paclitaxel Capsule; Drug: Encequidar tablet
- Stage 1: Oral Paclitaxel 205 mg/m2 + Encequidar (Experimental): A minimum of 20 subjects per group will be centrally randomized 1:1 to Oral Paclitaxel 165 mg/m2 + Encequidar 3 weeks of a 4-week cycle (3/4) or Oral Paclitaxel 205 mg/m2 (3/4) + Encequidar.
  Interventions: Drug: Paclitaxel Capsule; Drug: Encequidar tablet
- Stage 2: Oral Paclitaxel + Encequidar (Experimental)
  Interventions: Drug: Paclitaxel Capsule; Drug: Encequidar tablet
- Stage 2: IV Paclitaxel (Active Comparator)
  Interventions: Drug: IV Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel Capsule — Paclitaxel Capsule
  Arms: Stage 1: Oral Paclitaxel 165 mg/m2 + Encequidar; Stage 1: Oral Paclitaxel 205 mg/m2 + Encequidar; Stage 2: Oral Paclitaxel + Encequidar
Drug: IV Paclitaxel — IV Paclitaxel
  Arms: Stage 2: IV Paclitaxel
Drug: Encequidar tablet — Encequidar tablet
  Arms: Stage 1: Oral Paclitaxel 165 mg/m2 + Encequidar; Stage 1: Oral Paclitaxel 205 mg/m2 + Encequidar; Stage 2: Oral Paclitaxel + Encequidar

SUMMARY:
The current study is being conducted to find an optimal Oral Paclitaxel + Encequidar dose and regimen based on prior experience with oral paclitaxel (stage 1) and to compare that dose to an accepted dose and regimen of intravenous (IV) paclitaxel in subjects with metastatic breast cancer (stage 2).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. ≥18 years of age
3. Histologically or cytologically confirmed HER2 negative breast cancer for whom IV paclitaxel monotherapy has been recommended.
4. HER2 negative per American Society of Clinical Oncology (ASCO) College of American Pathologists (CAP) guideline. Subjects can be estrogen receptor/progesterone receptor (ER/PR) positive or negative per ASCO CAP guideline, but ER/PR and HER2 receptor status must be known.
5. Metastatic breast cancer with target lesions measurable by CT scan per RECIST v1.1 criteria confirmed by BICR
6. Adequate hematologic status as demonstrated by not requiring granulocyte colony stimulating factor (G CSF) or transfusion support within 30 days prior to randomization to achieve the following at screening:

   * Absolute neutrophil count (ANC) ≥1500/mm3
   * Platelet count ≥100,000/mm3
   * Hemoglobin ≥9 g/dL
7. Adequate liver function as demonstrated by:

   * Total bilirubin ≤upper limit of normal (ULN) unless the subject has Gilbert's disease, for which bilirubin must be ≤2.0 × ULN
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 × ULN
8. Adequate renal function as demonstrated by estimated glomerular filtration rate (eGFR) ≥60 mL/min
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
10. Life expectancy at least 6 months, in the judgment of the Investigator
11. Female subjects must be postmenopausal (≥12 months without menses) or surgically sterile (ie, by hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or must be using effective contraception (ie, non-hormonal intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of assigned study treatment.
12. Women of childbearing potential must have a negative screening serum pregnancy test and urine test within 4 days prior to start of dosing in the study and not be breast feeding.
13. Sexually active male subjects must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of investigational product (IP).

Exclusion Criteria:

1. Not recovered to ≤grade 1 toxicity from previous anticancer treatments or previous investigational product (IP) except alopecia
2. QTcF interval ≥470 msec at baseline
3. Relapsed less than 6 months following treatment with a taxane (paclitaxel or docetaxel) as part of anthracycline-based adjuvant chemotherapy or for metastatic disease
4. Known active central nervous system metastasis, including leptomeningeal involvement
5. Currently receiving other medications intended for the treatment of their malignancy
6. Received other IPs within 14 days or 5 half-lives of the first study dosing day, whichever is longer
7. Received biologics or monoclonal antibodies intended for the treatment of their malignancy within 30 days of the first study dosing day
8. Received radiation therapy within 2 weeks prior to signing informed consent or radiation therapy is planned within 6 months from the time of signing informed consent
9. Taking a medication known to be a moderate or strong cytochrome P450 (CYP) 3A4 inhibitor or inducer or neurokinin-1 receptor antagonist (NK-1) inhibitor within 14 days prior to start of dosing in the study
10. Taking a medication known to be a moderate or strong CYP2C8 inhibitor or inducer within 14 days prior to start of dosing in the study
11. Taking an oral medication with a narrow therapeutic index known to be a P-glycoprotein (P-gp) substrate within 24 hours prior to start of dosing in the study
12. Taking a medication known to be a P-gp inhibitor or inducer within 14 days prior to start of dosing in the study
13. Taking a medication known to be an organic anion transporting polypeptide 1B1/3 (OATP1B1/3) inhibitor
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, chronic pulmonary disease requiring oxygen, known bleeding disorders, or any concomitant illness or social situation that would limit compliance with study requirements
15. Major surgery to the upper GI tract, inability to take oral medication, or have a history of GI disease or other medical condition that, in the opinion of the Investigator may interfere with oral drug absorption
16. History of significant hypersensitivity-type reaction to paclitaxel or Cremophor EL that would contraindicate the use of IV paclitaxel
17. Known allergic reaction or intolerance to contrast media
18. Documented history of true systemic allergic reaction to 3 or more medications
19. Active hepatitis B (as evidenced by being HBsAg positive) or active hepatitis C (HCV-RNA positive) or cirrhosis of the liver
20. Known HIV infection
21. The Investigator believes that participation in this study would not be acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Confirmed Tumor Response | 6 months
  Confirmed tumor response based on BICR timepoint evaluations of CT scans using RECIST v1.1 criteria
Stage 2: Confirmed Tumor Response | 1 Year
  Confirmed tumor response based on BICR timepoint evaluations of CT scans using RECIST v1.1 criteria

IPD SHARING:
Plan to Share IPD: No